CLINICAL TRIAL: NCT04627714
Title: Physical and Moral Benefits of Adapted Fencing in Patients With Invasive Breast Cancer: Pilot Study of a Randomized Trial
Brief Title: Adapted Fencing in Breast Cancer: a Pilot Study
Acronym: RIPOSTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mathias POUSSEL, MD, PhD, Clinical Professor, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A01916-33
Record Dates: First submitted 2020-11-01; First posted 2020-11-13 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Breast Neoplasms
Keywords: Breast; Neoplams; adapted physical activity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Fencing (Experimental): patients of the "Early Fencing" arm will start adapted fencing practice (1h30/week) within 4 weeks after the breast surgery and for a duration of 3 months
  Interventions: Other: Adapted Physical Activity
- Delayed Fencing (Experimental): patients of the "Delayed Fencing" arm will start adapted fencing practice (1h30/week) 3 months after the breast surgery and for a duration of 3 months
  Interventions: Other: Adapted Physical Activity

INTERVENTIONS:
Other: Adapted Physical Activity — Intervention consists in 1h30/week of adapted fencing

SUMMARY:
Literature have shown the benefit of practicing regular physical activity during and after cancer treatment, particularly in terms of improving quality of life. The French Fencing Federation has thus developed an adapted physical activity program (Solution RIPOSTE) specially intended for patients with breast cancer. Adapted fencing sessions (saber) are thus offered to these patients in a perfectly secure context (i.e. compulsory medical-sports evaluation and trained fencing master). Since 2016, this RIPOSTE program has been implemented in several fencing halls in Lorraine. Our research project (controlled, randomized trial) aims to assess the impact of the practice of adapted fencing on the quality of life of patients, the functional capacities of the operated side (shoulder) and on the reduction of the sides effects of treatments. Our hypothesis is that such an adapted fencing program improves quality of life as well as functional abilities.

ELIGIBILITY:
Inclusion Criteria:

* Be a woman
* ≥ 18 years old.
* Have undergone unilateral breast surgery for primary invasive breast cancer
* Time between surgery and inclusion between 2 to 4 weeks after surgery
* Accept and be able to complete self-administered questionnaires
* Satisfy the prior medico-sports evaluation
* Be affiliated to a social security scheme or beneficiary of such a scheme
* Have received full information on the organization of the research and have signed their informed consent.

Exclusion Criteria:

* Presence of bone metastases, especially vertebral
* Presence of a contraindication to the practice of fencing during the medico-sports evaluation (post-surgery period that is too painful and / or requiring specific treatment in rehabilitation)
* Refusal to participate in the study
* Woman of childbearing age who does not have effective contraception.
* Persons referred to Articles L.1121-5, L.1121-7 and L. 1121-8 of the Public Health Code
* Pregnant woman, parturient or nursing mother
* Minor (non-emancipated)
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Person of full age unable to express consent
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric treatment under Articles L. 3212-1 and L. 3213-1.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline score of Quality of Life Questionnaire Core 30 (QLQ-C30) at 3 months. | Baseline (J0) and at 3 months (M3)
  Questionnaire. 30 items. minimum value = 30. Maximum value = 120. A high score means a worse outcome (i.e. poor quality of life)

SECONDARY OUTCOMES:
Change from baseline score of Disabilities of the Arm, Shoulder and Hand measurement tool (DASH) at 3 months | Baseline (J0) and at 3 months (M3)
  Questionnaire. 30 items. The score ranges from 0 (no disability) to 100 (most severe disability).
Change from baseline score of Multidimensional Fatigue Inventory (MFI-20) at 3 months | Baseline (J0) and at 3 months (M3)
  Questionnaire. 20 items. Minimal value = 20. Maximal value = 100. A high score means a worse outcome (i.e. high level of fatigue)
Change from baseline score of Hospital Anxiety and Depression Scale at 3 months. | Baseline (J0) and at 3 months (M3)
  Questionnaire. 14 items. The score ranges from 0 to 100. a high score means a worse outcome (i.e. high level of anxiety and depression)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias POUSSEL, MD, PhD, Principal Investigator — CHRU Nancy
Locations (3):
- France (3):
  - Hia Legouest, Metz
  - CHRU Nancy, Nancy
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omorou AY, Peiffert D, Rotonda C, Van Hoye A, Allado E, Hily O, Temperelli M, Chenuel B, Hornus-Dragne D, Poussel M. Adapted Fencing for Patients With Invasive Breast Cancer: The RIPOSTE Pilot Randomized Controlled Trial. Front Sports Act Living. 2022 Mar 29;4:786852. doi: 10.3389/fspor.2022.786852. eCollection 2022. PMID 35425895